CLINICAL TRIAL: NCT03952208
Title: Neurocognitive Dysfunction After Anesthesia in Patients With Recent Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Arnoley (Arney) S. Abcejo, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-006578
Record Dates: First submitted 2019-04-09; First posted 2019-05-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Concussion Group (Experimental): Subjects diagnosed with concussion defined as a clinician-diagnosed disease by the International Classification of Diseases (ICD)-10 due to a head injury with a Glasgow Coma Score ≥13 undergoing a planned surgery/anesthetic standard of care will undergo neurocognitive testing pre and post surgery/anesthetic.
  Interventions: Other: Neurocognitive Testing
- Matched Subjects Group (Experimental): Matched subjects without concussion undergoing a planned surgery/anesthetic standard of care, matching for procedural type, sex, age ± 2 years, and adherence to the exclusion criteria will undergo neurocognitive testing pre and post surgery/anesthetic.
  Interventions: Other: Neurocognitive Testing

INTERVENTIONS:
Other: Neurocognitive Testing — A comprehensive assessment of neuropsychometric measures to evaluate cognitive functioning.

SUMMARY:
Researchers are trying to determine if the impact of a concussion on the brain is affected by anesthesia and surgery.

DETAILED DESCRIPTION:
All subjects will complete pre and post procedure assessments prior to undergoing a planned surgery/anesthetic standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female >16 years of age with a recent concussion (<10 weeks) from planned procedure under anesthesia.

Exclusion Criteria:

* Neurologic history including history of severe cognitive disease, disorder, or delay, attention disorder, moderate to severe TBI history, neurovascular order or trauma.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Wide Range Achievement Test Fourth Edition, WRAT-4 | Pre-anesthetic to one week Post-anesthetic
  Change in WRAT-4

SECONDARY OUTCOMES:
Numeric Pain Scale 0-10 | Post-operatively to hospital discharge, up to 10 days.
  Difference in numeric pain scale between the concussion and non-concussion group. Patients verbally select a value that is in line with the intensity of pain they have experienced in the last 24 hours. Pain Scale is recorded "0" = no pain, "10" = the most pain imaginable.
Oral morphine equivalent of consumed opioids | Post-operatively to hospital discharge, up to 10 days.
  Difference of post-operative opioid use between the concussion and non-concussion group
Length of hospital stay | Post-operatively to hospital discharge, up to 30 days.
  Difference between the concussion and non-concussion group
Cognitive Deficits identified by NeuroPsychometric Cognitive Testing | Pre-anesthetic to one week Post-anesthetic
  Difference between the concussion and non-concussion group.
Sport Concussion Assessment Tool - 5th edition, SCAT-5 | Pre-anesthetic to one week Post-anesthetic
  The SCAT5 is a standardized tool for evaluating concussions designed for use by physicians and licensed medical professionals. Difference in SCAT5 scores between the concussion and non-concussion group. SCAT5 scores the number of symptoms (0-22) present and the severity of symptoms (0-132).

CONTACTS AND LOCATIONS:
Overall Officials: Arnoley S Abcejo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20450957